CLINICAL TRIAL: NCT02103374
Title: Evaluation of Benefit of Nebulized Bronchodilators at Home in Severe Chronic Obstructive Pulmonary Disease and Very Severe Steady State
Acronym: Nebuadom
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PHRN10-PD/Nebuadom; 2010-023743-14 (EudraCT Number); 2010-R38 (Other: CPP); A101466-30 (Other: Afssaps)
Record Dates: First submitted 2014-03-12; First posted 2014-04-03 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Severe Chronic Obstructive Pulmonary Disease
Keywords: weaned tobacco; Has not submitted an exacerbation in the past 3 months
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium; Terbutaline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atrovent + Bricanyl or Atrovent + Ventolin (Experimental): 3 daily inhalations of Atrovent mixture to form Bricanyl or Ventolin form Atrovent 0,5mg/1ml Bricanyl 5mg/2ml Ventolin 5mg/2,5ml
  Interventions: Drug: Atrovent + Bricanyl or Atrovent + Ventoline
- Placebo (Placebo Comparator): 1 capsule per day lactose (in addition to the standard optimized treatment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atrovent + Bricanyl or Atrovent + Ventoline — 3 daily inhalations of Atrovent mixture to form Bricanyl or Ventolin form during 48 weeks
  Arms: Atrovent + Bricanyl or Atrovent + Ventolin
Drug: Placebo — 1 capsule lactose during 48 weeks
  Arms: Placebo

SUMMARY:
Design studies of nebulization in COPD does not respond adequately to the clinically relevant question: the intervention of administering nebulized bronchodilators at home it is likely to make a profit, compared to the standard optimized treatment as defined by the recommendations of the SPLF, patients with severe COPD (stage III, FEV between 30% and 50% of the theoretical value) and very severe (stage IV, less than 30% of the theoretical value FEV)? The concept of profit in this context is based on criteria of dyspnea, quality of life, use of health system (exacerbations, hospitalizations, prescription of antibiotics and steroids ...).

ELIGIBILITY:
Inclusion Criteria:

* Adult
* COPD Patients stage 3 et 4
* Has not submitted an exacerbation in the 3 months preceding the pre-inclusion visit
* Weaned from tobacco for at least 6 months
* vaccinated against pneumococcal
* Have not been included in a pulmonary rehabilitation program during the 6 months preceding the screening visit inclusion
* Patient pre-included not showing exacerbation since the pre-inclusion visit

Exclusion Criteria:

* Patient under nebulizer or has been treated with nebulized bronchodilators at home over the last 6 months
* Patient with an indication of oxygen is expected in the coming year
* Progressive malignant disease known
* Patient under non-invasive ventilation (NIV) for less than 6 months or NIV provided in the following year
* Patient known to be colonized by Pseudomonas aeruginosa, A. xylosoxidans, Burkholderia cepacia or Stenotrophomonas maltophilia
* Patients with severe cardiovascular disease
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Score for quality of life, assessed by the questionnaire St Georges | Patients will be followed for the duration of their participation ie 48 weeks

SECONDARY OUTCOMES:
Score for quality of life, assessed by the questionnaire VQ11 | Patients will be followed for the duration of their participation ie 48 weeks
Dyspnea score according Medical Research Council | Patients will be followed for the duration of their participation ie 48 weeks
Prognostic Score Mortality assessed by the score BODE | Patients will be followed for the duration of their participation ie 48 weeks

OTHER OUTCOMES:
Number of exacerbations | Patients will be followed for the duration of their participation ie 48 weeks
Number of hospitalizations | Patients will be followed for the duration of their participation ie 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrice DIOT, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (13):
- France (13):
  - Service de Pneumologie, Amiens
  - Service de Pneumologie, Angers
  - Service de Pneumologie, Brest
  - Service de Pneumologie, Grenoble
  - Service de Pneumologie, Limoges
  - Service de Pneumologie, Nancy
  - Service de Pneumologie, Nantes
  - Service de Pneumologie, Orléans
  - Service de Pneumologie, Paris
  - Service de Pneumologie, Poitiers
  - Service de Pneumologie, Reims
  - Service de Pneumologie, Rouen
  - Service de Pneumologie, Tours